CLINICAL TRIAL: NCT06573229
Title: LIver FRAilty Management IN Cirrhosis (LIFRAMIN)
Acronym: LIFRAMIN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Rinninella Emanuele, MD, PhD, Researcher, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6409 - LIFRAMIN
Record Dates: First submitted 2024-08-26; First posted 2024-08-27 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Sarcopenia; Cirrhosis, Liver; Malnutrition; Protein
MeSH Terms: conditions — Sarcopenia; Liver Cirrhosis; Kwashiorkor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aminolife Plus (Experimental): Food supplement based on milk protein serum (Isolac Instant), acetyl-carnitine, hydroxy-methyl-butyrate, arginine, inositol, coenzyme Q10 and extracts of perilla, maca and mallow. Perilla supports the body's natural defences, maca has a tonic and metabolic support action and mallow has an emollient and soothing action (digestive system, urinary tract). Calcium, vitamin D and vitamin K2 complete the formulation. Calcium contributes to energy metabolism and is necessary for maintaining normal bones. Vitamin D modulates the immune system and contributes to regular muscle function. Vitamin aK2 contributes to proper blood clotting and maintenance of normal bones.
  Interventions: Dietary Supplement: Aminolife Plus by Piemme Pharmatech, Italy
- Placebo (Placebo Comparator): It is an inactive substance or treatment that has no therapeutic effect and is often used as a control in clinical trials.
  Interventions: Dietary Supplement: Aminolife Plus by Piemme Pharmatech, Italy

INTERVENTIONS:
Dietary Supplement: Aminolife Plus by Piemme Pharmatech, Italy — A nutritional supplement containing whey protein, vitamin D, carnitine, HMB, perilla, arginine, coenzyme Q10, inositol)

SUMMARY:
The goal of this clinical trial is to compare food for special medical purposes (Aminolife Plus, by Piemme Pharmatech) vs. placebo in improving muscle mass and function in a cohort of cirrhotic patients.

The main questions it aims to answer are:

* whether functional ability improves in cirrhotic-sarcopenic patients two months after taking the supplement compared with those not taking the supplement.
* whether weight, body mass index (BMI), lean mass, muscle mass, metabolically active mass, and phase angle as per bioimpedance analysis (BIA) in cirrhotic-sarcopenic patients increase two months after taking the supplement compared with those not taking the supplement.
* to assess quality-of-life indices in the two groups.
* to assess differences in groups in terms of plasma metabolite production in the two groups

This is a spontaneous, no PROFIT, pilot interventional study in the form of a randomized clinical trial (RCT), double-blind.

All patients will undergo simple sarcopenia risk identification questions (SARC-F test). All patients recognized to be at risk will be randomized to receive.

1. nutritional counseling according to guidelines + Aminolife plus 20 g/day (4 scoops) vs.
2. nutritional counseling according to guidelines + placebo 20 g/day (4 scoops) for a total of 60 days (2 months).

The manufacturing company will provide the product and placebo free of charge. Patients will undergo, at the first visit and at the follow-up visit anthropometric measurements and body composition assessment (by bioimpedance analysis).

In addition, 1 blood sample for metabolomic analysis will be taken at the same visits.

The study will last 12 months.

DETAILED DESCRIPTION:
patients will be randomly allocated within the two groups:

1. nutritional counselling according to guidelines + Aminolife plus 20 g/day (4 scoops) vs.
2. nutritional counselling according to guidelines + placebo 20 g/day (4 scoops)

The patients will be randomly allocated into two groups: the control group who will not take the treatment and the experimental group who will take the supplement. In detail, patients in the experimental group, in association with nutritional counselling, will take Aminolife plus 20 g/day (4 scoops) for two months (T0-T2).

Patients in the control group, in combination with nutritional counselling, will take placebo 20 g/day (4 scoops) for two months (T0-T2).

The division into the 2 groups will follow a block randomisation algorithm according to the Random Sorting procedure. The allocation sequence will be generated by means of the PASS2022 software.17 The allocation operator will be 'blinded' to the allocation group, just as the operator applying the treatment will not be involved in the evaluation of patients and results.

ELIGIBILITY:
Inclusion Criteria:

Patients affected by Liver cirrhosis

* at any stage of Child (A-B-C) with or without hepatocarcinoma
* SARC-F suggestive of risk of sarcopenia
* Age > 18 years
* Ability to perform Liver Frailty Index test
* Informed consent to participate in the study.

Exclusion Criteria:

* SARC-F not suggestive of sarcopenia
* inability to perform Liver Frailty Index test
* absence of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-08-02 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Improved functional capacity (Liver Frailty Index) | 12 months
  Improved functional capacity in cirrhotic-sarcopenic patients, assessed by using the Liver Frailty Index test, which has already been validated in the literature and includes 3 continuous parameters (Handgrip strenght test, Chair Stand Test and Balance test).

SECONDARY OUTCOMES:
Improved anthropometric and bioelectrical values and comparing the two | 12 months
  Differences between the two groups in weight, body mass index (BMI), lean mass, muscle mass, metabolically active mass, and phase angle, as per bioimpedance analysis (BIA);
Improved QoL | 12 months
  Differences in quality of life indices (QLQ-C30, QLQ-CR29, QLQ-CAX24, QLQ-PRT20) between the two groups.
Differences in terms of plasmatic metabolites | 12 months
  Differences between the 2 intervention groups in terms of plasma metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Rinninella, PI, Principal Investigator — Fondazione Policlinico Gemelli, Rome
Locations (1):
- Emanuele Rinninella, Rome, Italy